CLINICAL TRIAL: NCT02985112
Title: INTegrated Assessment of intERmediate Coronary Stenoses by Fractional Flow rEserve (FFR) and Near-infraREd Spectroscopy (NIRS).
Acronym: INTERFERE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: S.M. Misericordia Hospital (Other)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Principal Investigator, Andrea Picchi, Principal Investigator, S.M. Misericordia Hospital
Other Study IDs: USL9-2015-007-NIRS
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Borderline Coronary Stenoses Assessment, Fractional Flow Reserve, Plaque Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (2):
- Patients with FFR > 0.80: Group of patients with physiologically non-significant coronary stenoses who will not undergo coronary revascularization
  Interventions: Device: FFR and IVUS-NIRS
- Patients with FFR < 0.80: Group of patients with physiologically significant coronary stenoses who will undergo coronary revascularization
  Interventions: Device: FFR and IVUS-NIRS

INTERVENTIONS:
Device: FFR and IVUS-NIRS

SUMMARY:
Revascularization of borderline coronary stenoses (40-70%) is usually driven by fractional flow reserve (FFR) which expresses the physiological significance of a lesion and tells the operator whether PCI may reduce the rate of adverse events as compared to medical therapy. Coronary stenoses with FFR value < 0.80 are indeed associated with a higher rate of adverse event and requires coronary revascularization whereas lesions with FFR > 0.80 show an excellent prognosis which cannot be improved by coronary stenting. Such a predictive value of FFR is theoretically based only on the degree of myocardial ischemia downstream from a given coronary stenosis: however, also plaque composition may play a crucial role in triggering future events especially in patients affected by acute coronary syndrome. Differences in plaque composition between FFR-positive and FFR negative lesions have never been assessed. Intracoronary Near-InfraRed Spectroscopy (NIRS) identifies lipid rich plaques that can potentially cause acute events. The aim of this study is to compare the lipid content expressed by LCBI (Lipid Core Burden Index) between functionally significant (FFR < 0.80) and non-significant (FFR > 0.80) stenoses in patients undergoing coronary angiography because of stable CAD and non-ST elevation acute coronary syndromes. This is an observational, prospective, multicentric study where we plan to collect 150 coronary lesions.

DETAILED DESCRIPTION:
Background Objective of percutaneous coronary intervention (PCI) is the treatment of angiographically significant coronary stenoses in patients affected by stable or unstable coronary syndromes 1. When we face an intermediate stenosis (percentage diameter stenosis between 40% and 70%), revascularization is guided by the presence of inducible myocardial ischemia, detected by non - invasive stress tests or by assessment of fractional flow reserve (FFR). FFR is an index of the physiological significance of a coronary stenosis and is defined as the ratio of maximal blood flow in a stenotic artery to normal maximal flow. An FFR value of 0.80 or less identifies ischemia-causing coronary stenoses with an accuracy of more than 90%. FFR is a very accurate tool to identify functionally significant stenoses and to predict cardiovascular events in patients with stable coronary artery disease (CAD) and solid evidences demonstrate that PCI of lesions with FFR > 0.80 can be safely deferred (incidence of MACE < 1% with medical treatment only). Conversely, stenoses with an FFR <0.80 have a poor prognosis and require treatment by PCI 2-4. The afore-mentioned indications come from studies that mainly involved patients affected by stable CAD, but the role of FFR in the setting of acute coronary sindrome (ACS) is less clear. Hakeem et al. have recently shown that deferring percutaneous coronary intervention on the basis of non-ischemic FFR in patients with an initial presentation of ACS is associated with significantly worse outcomes than stable patients5.

FFR indeed has the ability to identify vessels with reduced coronary flow, but cannot detect atherosclerotic plaques with unstable features, which may present without flow limitation (FFR > 0.80) but can cause acute coronary events 6, 7. Since the prevalence of features of plaque instability (plaque volume > 70%, minimum luminal area <4 mm2, presence of a "thin cap fibroatheroma") increase with the increase of the severity of the stenosis, the decision of performing PCI for stenoses of clear angiographic severity seems rational and supported by solid evidence 8. Conversely, delaying PCI of intermediate stenoses on the basis of a negative FFR can be problematic, particularly in patients with ACS, where the only functional evaluation with FFR may not be sufficient in the presence of unstable plaques.

Differences in plaque composition between physiologically significant vs non-significant lesions have never been assessed in either stable and ACS patients.

Intracoronary Near-InfraRed Spectroscopy (NIRS) identifies lipid-rich plaques (LRP) with high sensibility and specificity. The technique, validated on autopsy specimens, is an effective tool to detect LRP in vivo, identifying those coronary atheromas that can potentially cause acute events 9. The NIRS system consists of a 3.2-F rapid exchange catheter (InfraReDx, Burlington,Massachusetts), a pullback and rotation device, and a console. The measurement of the probability of LRP for each scanned arterial segment is displayed as a map, with the x-axis indicating the pullback position in millimeters and the y-axis the circumferential position of the measurement in degrees. The algorithm displays the probability of lipid content at the interrogation site by using a false color scale from red (low probability) to yellow (high probability). The entire display is termed a "chemogram". Pixels containing insufficient informations are displayed as black. The ratio between the number of yellow pixels to the whole number of pixels except the black ones, multiplied by one - thousand, is the "Lipid Core Burden Index (LCBI)" of the analyzed artery segment. A value of LCBImax > 400 identifies a high lipid content in a given segment. In an autopsy study conducted on human aortic specimens, the technique reached 90% sensibility and 93 % specificity in the detection of lipid rich plaques9, opening new horizons in terms of risk stratification and therapy10-15. To provide a quantitative target suitable for algorithm construction and validation, a lipid core plaque of interest was defined as a fibroatheroma with a lipid core > 60° in circumferential extent, >200 µm thick, with a fibrous cap having a mean thickness < 450 µm16.

Aim of the study

* To compare lipid content expressed by LCBImax value between functionally significant (FFR < 0.80) and non-significant (FFR > 0.80) stenoses in patients undergoing coronary angiography because of stable CAD and non-ST elevation acute coronary syndromes.
* To evaluate the correlation between functional significance (expressed by FFR value) and lipid content (expressed by LCBImax value) of coronary lesions in patients undergoing coronary angiography because of stable CAD and non-ST elevation acute coronary syndromes.

Design of the study This is an observational, prospective, multicentric study: at present time, two centers (Misericordia Hospital, Grosseto and San Giovanni Hospital, Rome) are going to take part in the study.

Subjects undergoing coronary angiography for stable CAD and non-ST-segment elevation acute myocardial infarction (NSTEMI) and unstable angina will be enrolled. Patients included must have evidence of at least one angiographically borderline stenosis (≥ 40, <70% by Quantitative Coronary Angiography, QCA) with normal antegrade flow (TIMI 3). The index lesion will be evaluated by FFR; afterwards, plaque composition and lesion characteristics will be evaluated by IVUS - NIRS. PCI will be performed according to current guidelines on myocardial revascularization1.

Patients with hemodynamic instability, ST-segment-elevation myocardial infarction, known allergy to antiplatelet or anticoagulant drugs, history of previous CABG, significant left main disease, life expectancy < 1 year, severe renal failure, malignancy, scheduled valve surgery, inability to provide informed consent, known bronchial asthma, age < 18 will be excluded.

Endpoints

* Primary endpoint: percentage of coronary plaques with LCBImax > 400 in lesions with FFR > 0.80 vs lesions with FFR < 0.80. .
* Secondary endpoints: 1) lipid content expressed as LCBImax (mean ± SD) in lesions with FFR > 0.80 vs lesions with FFR < 0.80. 2) Correlation between lipid content (as LCBI max), and functional significance (as FFR) of the index lesion.

Sample size The sample size will be calculated to demonstrate a decrease in the primary end point (percentage of coronary plaques with LCBImax > 400) from 36% in FFR positive lesions to 18% in FFR negative lesions, as inferred by previous findings showing a 36% vs 18% prevalence of thin cap fibroatheroma in lesions with a >70% vs <70% diameter stenosis17. Using chi-square test for 2 x 2 tables and a 1-sided alpha value of 0.05, a sample of 150 lesions will provide the study 80% power to meet the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing coronary angiography for stable CAD and non-ST-segment elevation acute myocardial infarction (NSTEMI) and unstable angina will be enrolled. Patients included must have evidence of at least one angiographically borderline stenosis (≥ 40, <70% by Quantitative Coronary Angiography, QCA) with normal antegrade flow (TIMI 3). The index lesion will be evaluated by FFR; afterwards, plaque composition and lesion characteristics will be evaluated by IVUS - NIRS. PCI will be performed according to current guidelines on myocardial revascularization1.

Exclusion Criteria:

* Patients with hemodynamic instability, ST-segment-elevation myocardial infarction, known allergy to antiplatelet or anticoagulant drugs, history of previous CABG, significant left main disease, life expectancy < 1 year, severe renal failure, malignancy, scheduled valve surgery, inability to provide informed consent, known bronchial asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing coronary angiography for stable CAD and non-ST-segment elevation acute myocardial infarction (NSTEMI) and unstable angina will be enrolled. Patients included must have evidence of at least one angiographically borderline stenosis (≥ 40, <70% by Quantitative Coronary Angiography, QCA) with normal antegrade flow (TIMI 3). The index lesion will be evaluated by FFR; afterwards, plaque composition and lesion characteristics will be evaluated by IVUS - NIRS. PCI will be performed according to current guidelines on myocardial revascularization1.
  Patients with hemodynamic instability, ST-segment-elevation myocardial infarction, known allergy to antiplatelet or anticoagulant drugs, history of previous CABG, significant left main disease, life expectancy < 1 year, severe renal failure, malignancy, scheduled valve surgery, inability to provide informed consent, known bronchial asthma, age < 18 will be excluded.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of coronary plaques with LCBImax > 400 in lesions with FFR > 0.80 vs lesions with FFR < 0.80. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Unit, Misericordia Hospital, Grosseto, Italy, Italy

REFERENCES:
- [Derived] Picchi A, Campo G, Misuraca L, Baratta P, Biancofiore A, Calabria P, Massoni A, Limbruno U. INTegrated Assessment of intERmediate Coronary Stenoses by Fractional Flow rEserve and Near-infraREd Spectroscopy: The INTERFERE Study. J Clin Med. 2025 Sep 25;14(19):6769. doi: 10.3390/jcm14196769. PMID 41095849